CLINICAL TRIAL: NCT04328298
Title: French Register Of Patients With Hemopathy Eligible For CAR-T Cell Treatment (DESCAR-T)
Status: Recruiting | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Gilead Sciences (Industry); Novartis (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: DESCAR-T
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hematopathology Eligible or CAR-t Cell Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a registry including prospective and retrospective data on all patients who have been presented in a Multidisciplinary tumor board or RCP to be eligible for CAR-T cell treatment.

ELIGIBILITY:
Inclusion Criteria:

Retrospective inclusion :

* Patient treated with CAR-T from 1 July 2018 under temporary authorization (ATU) or covered by French health insurance system (under post-ATU or MA) in a qualified center before activation of this register in this center
* If the patient is alive, the patient has been informed of the collection and use of their data, and the patient has not opposed this use. If the patient has died, the patient did not opposed the use of their data while alive

Prospective inclusion :

* Patient eligible for a treatment with CAR-T for an hematological malignancy which is covered by French health insurance (for ATUs / post-ATUs or MA), or as part of a clinical trial with the same indication, after the activation of this register in this center.
* Patient whose CAR-T indication has been validated during a multidisciplinary tumor board (RCP) of a qualified center, according to the ministerial order of 8 August 2019
* Patient deemed eligible for a treatment with CAR-T after a medical exam performed in a qualified center according to the ministerial order of 8 August 2019
* If the patient is alive, the patient has been informed of the collection and use of their data, and the patient has not opposed this use. If the patient has died, the patient did not opposed the use of their data while alive.

Exclusion Criteria Patient not registered with the social security in France

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient eligible for a treatment with CAR-T for an hematological malignancy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2038-12-19 (Estimated); Study Completion 2038-12-19 (Estimated)

PRIMARY OUTCOMES:
overall survival from eligibility | 15 years
Overall survival from administration | 15 years
complete response rate | 15 years
Progression free survival | 15 years
Duration of response | 15 years
Delays between patient eligibility and CAR-T treatment | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, Pr, Principal Investigator — Institut Curie; Roch HOUOT, Pr, Principal Investigator — CHU Pontchaillou
Locations (36):
- France (36):
  - CHU d'Amiens - Hôpital Sud, Amiens
  - CHU Angers, Angers
  - CHRU Besançon - Hôpital Minjoz, Besançon
  - CHU de Brest - Hôpital du Morvan, Brest
  - Institut d'Hématologie de Basse Normandie, Caen
  - CHU d'Estaing, Clermont-Ferrand
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, La Tronche
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut d'Hématologie et d'Oncologie Pédiatrique (IHOP), Lyon
  - Hôpital de la Timone, Marseille
  - Institut Paoli Calmette, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU de Nice, Nice
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital La Pitié Salpêtrière, Paris
  - APHP - Hôpital Necker, Paris
  - APHP - Hôpital Saint Antoine, Paris
  - APHP - Hôpital Saint Louis, Paris
  - APHP - Hôpital Universitaire Robert Debré, Paris
  - Centre Francois Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de la Milétrie - CHU de Poitiers, Poitiers
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU de Rouen Normandie, Rouen
  - Institut de Cancérologie Hématologie Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - ICANS (Institut de Cancérologie Strasbourg Europe), Strasbourg
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
  - CHU Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cayla S, Karlin L, Lambert J, Lazareth A, Talbot A, Mohty M, Malard F, Petillon MO, Manier S, Yakoub-Agha I, Caillot D, Lafon I, Leleu X, Moya N, Royer B, Schiano de Colella JM, Brisou G, Touzeau C, Perrot A, Bories P, Vincent L, Guedon H, Decaux O, Ferment B, Houot R, Le Gouill S, Bigot N, Facon T, Corre J, Avet-Loiseau H, Moreau P, Arnulf B. Poor Outcomes with BCMA-targeting bispecific antibodies following early relapse from ide-cel: a real-world French study. Blood Adv. 2025 Sep 18:bloodadvances.2025017597. doi: 10.1182/bloodadvances.2025017597. Online ahead of print. PMID 40966637
- [Derived] Sesques P, Kirkwood AA, Kwon M, Rejeski K, Jain MD, Di Blasi R, Brisou G, Gros FX, le Bras F, Bories P, Choquet S, Rubio MT, Iacoboni G, O'Reilly M, Casasnovas RO, Bay JO, Mohty M, Joris M, Abraham J, Castilla Llorente C, Loschi M, Carras S, Chauchet A, La Rochelle LD, Hermine O, Guidez S, Cony-Makhoul P, Fogarty P, Le Gouill S, Morschhauser F, Gastinne T, Cartron G, Subklewe M, Locke FL, Sanderson R, Barba P, Houot R, Bachy E. Novel prognostic scoring systems for severe CRS and ICANS after anti-CD19 CAR T cells in large B-cell lymphoma. J Hematol Oncol. 2024 Aug 6;17(1):61. doi: 10.1186/s13045-024-01579-w. PMID 39107847
- [Derived] Bachy E, Le Gouill S, Di Blasi R, Sesques P, Manson G, Cartron G, Beauvais D, Roulin L, Gros FX, Rubio MT, Bories P, Bay JO, Llorente CC, Choquet S, Casasnovas RO, Mohty M, Guidez S, Joris M, Loschi M, Carras S, Abraham J, Chauchet A, Drieu La Rochelle L, Deau-Fischer B, Hermine O, Gastinne T, Tudesq JJ, Gat E, Broussais F, Thieblemont C, Houot R, Morschhauser F. A real-world comparison of tisagenlecleucel and axicabtagene ciloleucel CAR T cells in relapsed or refractory diffuse large B cell lymphoma. Nat Med. 2022 Oct;28(10):2145-2154. doi: 10.1038/s41591-022-01969-y. Epub 2022 Sep 22. PMID 36138152